CLINICAL TRIAL: NCT02608229
Title: Phase Ib Study of BVD-523 Plus Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Brief Title: BVD-523 Plus Nab-paclitaxel and Gemcitabine in Patients With Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adverse events
Sponsor: Washington University School of Medicine (Other)
Collaborators: BioMed Valley Discoveries, Inc (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201601098; 5P50CA196510-02 (NIH)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2020-05-01 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer; Cancer of Pancreas; Cancer of the Pancreas; Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ulixertinib; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine (Experimental): * Treatment will be given in a 28-day cycle.
  * BVD-523 600 mg on a twice daily basis (at approximately 12-hour intervals).
  * BVD-523 at 600 mg twice daily on its own for two weeks before initiating Cycle 1 treatment with gemcitabine and nab-paclitaxel.
  * Nab-paclitaxel 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30-40 minutes.
  * Gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30 minutes.
  * Mandatory biopsy at baseline and baseline at end of 2 week BVD-523 lead in.
  Interventions: Drug: BVD-523; Drug: Nab-paclitaxel; Drug: Gemcitabine; Procedure: Tumor biopsy
- Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine (Experimental): * Treatment will be given in a 28-day cycle.
  * First 2 patients enrolled: BVD-523 600 mg on a twice daily basis (at approximately 12-hour intervals), nab-paclitaxel 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30-40 minutes, and gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30 minutes
  * Remaining 6 patients enrolled: BVD-523 450 mg on a twice daily basis (at approximately 12-hour intervals), nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30-40 minutes, and gemcitabine 800 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30 minutes
  * Mandatory biopsy at baseline and at end of cycle 2 (if deemed safe for participant and feasible to obtain)
  Interventions: Drug: BVD-523; Drug: Nab-paclitaxel; Drug: Gemcitabine; Procedure: Tumor biopsy

INTERVENTIONS:
Drug: BVD-523
Drug: Nab-paclitaxel
  Other Names: Abraxane; Paclitaxel Albumin-stabilized Nanoparticle Formulation
Drug: Gemcitabine
  Other Names: Gemcitabine hydrochloride; Gemzar
Procedure: Tumor biopsy

SUMMARY:
In light of the central role of extracellular signal-regulated kinases (ERK) in pancreatic cancer, the investigators propose a phase I study to evaluate the ERK inhibitor BVD-523 at the recommended phase 2 dose in combination with nab-paclitaxel plus gemcitabine in patients with newly diagnosed metastatic pancreatic cancer. The primary endpoint will be maximum tolerated dose (MTD) or RP2D and safety. The secondary endpoints include safety, response rate, biochemical response, progression-free survival (PFS) and overall survival (OS). The exploratory endpoints include the assessing the impact of BVD-523 on the MEK/ERK pathway and other major pathway pertain to pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed newly diagnosed treatment-naïve metastatic adenocarcinoma of the pancreas with metastatic disease diagnosed no more than 6 weeks prior to enrollment. Patients with advanced pancreatic cancer progressed on 5-FU (or capecitabine) based regimen will be allowed in the expansion cohort.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* Life expectancy > 3 months.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN, unless there are liver metastases in which case AST and ALT ≤ 5.0 x IULN
  * Creatinine ≤ 1.5 x IULN OR GFR of ≥ 50 mL/min
  * Cardiac function ≥ ILLN, e.g., LVEF of > 50% as assessed by MUGA or ECHO, QTc < 470 ms
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for three months following study discontinuation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Current use or anticipated need for alternative, holistic, naturopathic, or botanical formulations used for the purpose of cancer treatment.
* A history of other malignancy with the exception of those treated with curative intent with no evidence of disease for 2 years.
* Currently receiving any other investigational agents.
* Known brain metastases or CNS involvement.
* Significant ascites that require therapeutic paracentesis.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to BVD-523, gemcitabine, nab-paclitaxel, or other agents used in the study.
* Neuropathy ≥ grade 2.
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* History of interstitial lung disease or pneumonitis.
* Concurrent therapy with drugs known to be strong inhibitors of CYP1A2, CYP2D6, and CYP3A4, or strong inducers of CYP3A4 (see Appendix B).
* Gastrointestinal condition which could impair absorption of BVD-523 or inability to ingest BVD-523.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of study entry.
* Known HIV-positivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grierson PM, Tan B, Pedersen KS, Park H, Suresh R, Amin MA, Trikalinos NA, Knoerzer D, Kreider B, Reddy A, Liu J, Der CJ, Wang-Gillam A, Lim KH. Phase Ib Study of Ulixertinib Plus Gemcitabine and Nab-Paclitaxel in Patients with Metastatic Pancreatic Adenocarcinoma. Oncologist. 2023 Feb 8;28(2):e115-e123. doi: 10.1093/oncolo/oyac237. PMID 36427020
- [Derived] Germann UA, Furey BF, Markland W, Hoover RR, Aronov AM, Roix JJ, Hale M, Boucher DM, Sorrell DA, Martinez-Botella G, Fitzgibbon M, Shapiro P, Wick MJ, Samadani R, Meshaw K, Groover A, DeCrescenzo G, Namchuk M, Emery CM, Saha S, Welsch DJ. Targeting the MAPK Signaling Pathway in Cancer: Promising Preclinical Activity with the Novel Selective ERK1/2 Inhibitor BVD-523 (Ulixertinib). Mol Cancer Ther. 2017 Nov;16(11):2351-2363. doi: 10.1158/1535-7163.MCT-17-0456. Epub 2017 Sep 22. PMID 28939558
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/06/2016 and closed to participant enrollment on 08/19/2019.
Period: Overall Study
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Started | 10 | 8
600 mg BVD-523 | 10 | 2
450 mg BVD-523 | 0 | 6
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Median (Full Range); unit: years] | 65.5 [55 to 74] | 61.5 [37 to 78] | 63.5 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BVD-523
Description: -The maximum tolerated dose (MTD) is defined as the Dose Level 1 if 0 or 1 dose-limiting toxicities (DLTs) are seen in patients at that dose level or Dose Level -1 if 2+ DLTs are seen in Dose Level 1 but only 0 or 1 DLTs are seen in patients at Dose Level -1.
Time Frame: Completion of cycle 1 for all dose de-escalation patients (1.8 years), the first cycle is 28 days for each individual patient
Population: -The MTD was not determined by DLTs in Dose De-escalation. 2 patients in Dose Expansion were treated at 600 mg but due to poor performance (inability to complete Cycle 1) the principal investigator felt it was reasonable to treat the remaining patients with 450 mg BVD-523 twice daily in the dose expansion portion of the study.
Measure: Number; unit: mg
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 10 | 0
mg | 450 |

2. Secondary Outcome: Safety and Toxicity Profile of Treatment Regimen as Measured by Grade and Frequency of Adverse Events
Description: -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Time Frame: 30 days after completion of treatment (median time was 67.5 days)
Measure: Count of Participants; unit: Participants
Groups:
- 600 mg BVD-523/Nab-paclitaxel/Gemcitabine: * Treatment will be given in a 28-day cycle.
  * All patients who received 600 mg BVD-523 on a twice daily basis (at approximately 12-hour intervals) are included in this group
  * Nab-paclitaxel 125 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30-40 minutes.
  * Gemcitabine 1000 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30 minutes.
- 450 mg BVD-523/Nab-paclitaxel/Gemcitabine: * Treatment will be given in a 28-day cycle.
  * All patients who received 450 mg BVD-523 on a twice daily basis (at approximately 12-hour intervals) are included in this group
  * Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30-40 minutes.
  * Gemcitabine 800 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle over the course of 30 minutes.
Arm/Group | 600 mg BVD-523/Nab-paclitaxel/Gemcitabine | 450 mg BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 12 | 6
Participants
  Grade 1/2 Hearing Impaired | 1 | 0
  Grade 1/2 blurred vision | 3 | 0
  Grade 3 abdominal infection | 1 | 0
  Grade 1/2 constipation | 5 | 2
  Grade 1/2 diarrhea | 5 | 4
  Grade 3 diarrhea | 2 | 0
  Grade 1/2 dry mouth | 2 | 0
  Grade 1/2 dyspepsia | 1 | 1
  Grade 1/2 flatulence | 1 | 0
  Grade 1/2 gastrointestinal pain | 1 | 0
  Grade 1/2 mucositis oral | 2 | 2
  Grade 1/2 nausea | 5 | 1
  Grade 3 nausea | 1 | 1
  Grade 1/2 taste change | 1 | 0
  Grade 1/2 vomiting | 0 | 1
  Grade 3 vomiting | 2 | 1
  Grade 1/2 acute kidney injury | 1 | 0
  Grade 3 lower GI hemorrhage | 1 | 0
  Grade 1/2 chills | 3 | 1
  Grade 1/2 edema limbs | 3 | 1
  Grade 1/2 edema trunk | 1 | 0
  Grade 1/2 fatigue | 3 | 2
  Grade 1/2 fever | 5 | 2
  Grade 1/2 thrush | 1 | 1
  Grade 5 death due to disease progression | 1 | 1
  Grade 1/2 alanine aminotransferase increased | 2 | 0
  Grade 1/2 alkaline phosphtase | 2 | 0
  Grade 4 blood bilirubin increased | 1 | 0
  Grade 3/4 neutrophil count decreased | 3 | 1
  Grade 3 platelet count decreased | 1 | 1
  Grade 1/2 lymphocyte count | 1 | 0
  Grade 1/2 white blood cell count decreased | 2 | 0
  Grade 1/2 hypercalcemia | 2 | 0
  Grade 1/2 hyperglycemia | 1 | 0
  Grade 1/2 hyperkalemia | 2 | 0
  Grade 1/2 hypoalbuminemia | 1 | 0
  Grade 1/2 hypocalcemia | 1 | 0
  Grade 1/2 dehydration | 1 | 1
  Grade 1/2 arthralgia | 4 | 1
  Grade 1/2 back pain | 2 | 0
  Grade 1/2 dizziness | 4 | 1
  Grade 1/2 headache | 3 | 0
  Grade 1/2 peripheral sensory neuropathy | 5 | 0
  Grade 1/2 numbness | 1 | 0
  Grade 1/2 insomnia | 2 | 1
  Grade 1/2 anxiety | 1 | 1
  Grade 1/2 cough | 1 | 1
  Grade 1/2 dyspnea | 2 | 0
  Grade 1/2 epistaxis | 1 | 0
  Grade 5 adult respiratory distress syndrome | 1 | 0
  Grade 1/2 alopecia | 5 | 3
  Grade 1/2 rash acneiform | 3 | 4
  Grade 3 rash acneiform | 2 | 0
  Grade 1/2 rash maculo-papular | 4 | 0
  Grade 1/2 sweating | 1 | 0
  Grade 1 scalp sun burned | 1 | 0
  Grade 1/2 hypertension | 3 | 0
  Grade 3 hypertension | 1 | 0
  Grade 1/2 hyperhydrosis | 0 | 1
  Grade 1/2 pruritus | 0 | 1
  Grade 1/2 myalgia | 0 | 1
  Grade 1/2 blood in stool | 0 | 1
  Grade 1/2 anorexia | 3 | 1
  Grade 3 anorexia | 0 | 1
  Grade 1/2 abdominal pain | 2 | 2
  Grade 3 abdominal pain | 0 | 1
  Grade 3 portal vein thrombosis | 0 | 1
  Grade 3 lung infection | 0 | 1
  Grade 1/2 anemia | 3 | 1
  Grade 3 anemia | 0 | 1

3. Secondary Outcome: Response Rate
Description: * Response rate is the percentage of participants with best response of complete response or partial response per RECIST 1.1
  * Complete response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Disappearance of all non-target lesions and normalization of tumor marker level.
  * Partial response (PR): at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through completion of treatment (median time was 37.5 days)
Population: Participants who did not have a follow-up CT scan were excluded from this outcome measure. The 2 participants analyzed in the Dose Expansion arm received 450 mg of BVD-523.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 5 | 2
Participants | 2 | 0

4. Secondary Outcome: Biochemical Response of Treatment Regimen
Description: -The biochemical response (BR) is defined as more than 50% of decrease from baseline CA 19-9
Time Frame: Through completion of treatment (median time was 37.5 days)
Population: -Participants with normal CA19-9 levels at baseline were excluded from this outcome measure and those who did not have an additional CA19-9 level drawn after baseline. Of the 5 participants analyzed in Dose Expansion Arm, 1 received 600 mg BVD-523 and 4 participants received 450 mg BVD-523.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 7 | 5
Participants | 3 | 1

5. Secondary Outcome: Time to Tumor Progression (TTP)
Description: * Time to tumor progression is defined as the days from start of treatment until progressive disease.
  * Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Up to 2 years
Population: Participants who did not have a follow-up CT scan were excluded from this outcome measure. The 2 participants analyzed in the Dose Expansion Arm received 450 mg BVD-523.
Measure: Median (Full Range); unit: days
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 5 | 2
days | 85 [63 to 243] | 39.5 [30 to 49]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: * Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Patients alive without progression or lost to follow-up are censored.
Time Frame: Up to 2 years
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | Dose De-escalation: BVD-523/Nab-paclitaxel/Gemcitabine | Dose Expansion: BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 5 | 2
days | 85 [63 to 243] | 39.5 [30 to 49]

7. Secondary Outcome: Overall Survival (OS)
Description: -OS is defined as the days from the date of treatment start and death from any cause. Participants alive or lost to follow-up are censored.
Time Frame: Up to 2 years
Population: Participants were not considered evaluable for this outcome measure if they were not evaluable for dose-limiting toxicities per protocol and any participants that were alive were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 600 mg BVD-523/Nab-paclitaxel/Gemcitabine | 450 mg BVD-523/Nab-paclitaxel/Gemcitabine
Number analyzed (Participants) | 6 | 6
months | 13.8 [10.7 to 22.8] | 5.7 [1.1 to NA] — There were too few participants to provide upper estimate on the 95% confidence interval.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of study treatment until 30 days following completion of study treatment. Median length of follow-up for adverse events was 67.5 days.
Arm/Group | 600 mg BVD-523/Nab-paclitaxel/Gemcitabine | 450 mg BVD-523/Nab-paclitaxel/Gemcitabine
All-Cause Mortality (participants affected / at risk) | 11/12 | 5/6
Serious Adverse Events (participants affected / at risk) | 8/12 | 4/6
Other Adverse Events (participants affected / at risk) | 12/12 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg BVD-523/Nab-paclitaxel/Gemcitabine (N=12) | 450 mg BVD-523/Nab-paclitaxel/Gemcitabine (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Lower GI hemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Death due to disease progression (General disorders) | 1 | 1
Fever (General disorders) | 5 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg BVD-523/Nab-paclitaxel/Gemcitabine (N=12) | 450 mg BVD-523/Nab-paclitaxel/Gemcitabine (N=6)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Blurred vision (Eye disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 6 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 5 | 1
Taste change (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Chills (General disorders) | 3 | 1
Edema limb (General disorders) | 3 | 1
Edema trunk (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
Fever (General disorders) | 0 | 2
Thrush (General disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0
Numbness (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp sun burned (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 4 | 0
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Blood in stool (Gastrointestinal disorders) | 0 | 1
Portal vein thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02608229/Prot_SAP_001.pdf